CLINICAL TRIAL: NCT00201656
Title: Removal Versus Retention of Cervical Cerclage in Preterm Premature Rupture of Membranes-A Multicenter Randomized Clinical Trial
Brief Title: Removal Versus Retention of Cerclage in Preterm Premature Rupture of Membranes (PPROM)
Acronym: PROMCerclage
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This trial was terminated following a futility analysis confirming futility of continuing the study
Sponsor: Obstetrix Medical Group (Industry)
Responsible Party: Sponsor
Organization: Pediatrix (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBX0002; OBX0002 (Other: Obstetrix CREQ Protocol Number)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Fetal Membranes, Premature Rupture
Keywords: PPROM; Cerclage; Preterm Premature Rupture of the Membranes with Cerclage
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Retention of Cerclage (Active Comparator): Group one = Subject whose Cerclage is retained after randomization.
  Interventions: Procedure: Retention of Cerclage; Procedure: Removal vs. Retention of Cervical Cerclage
- 2 - Removal of Cerclage (Active Comparator): Group 2 = Subjects who will have cerclage removed after randomization
  Interventions: Procedure: Removal of Cerclage; Procedure: Removal vs. Retention of Cervical Cerclage

INTERVENTIONS:
Procedure: Retention of Cerclage — Retain Cerclage until clinical removal is indicated by protocol
  Arms: 1 Retention of Cerclage
Procedure: Removal of Cerclage — Immediate removal of Cerclage following randomization
  Arms: 2 - Removal of Cerclage
Procedure: Removal vs. Retention of Cervical Cerclage — Immediate removal of cerclage following randomization vs. retention of cerclage until labor, chorioamnionitis, or fetal distress
  Other Names: McDonald or Shirodkar Cerclage

SUMMARY:
The purpose of this study is to determine whether retention of cervical cerclage after PPROM improves latency (without a significant increase in chorioamnionitis) and lessens neonatal morbidity.

DETAILED DESCRIPTION:
The placement of cervical cerclage is standard of care for women who experience incompetent cervix. Treadwell et al, published the largest retrospective review of 482 patients receiving cerclage (364 elective and 118 emergent). They found premature rupture of membranes (PROM) in 38% of the subjects with 9% delivering <27 weeks. Preterm birth is the cause of at least 75% of neonatal deaths that are not due to congenital malformations. The question of whether to remove cerclage after preterm premature rupture of membranes (PPROM) is one of the unresolved controversies in obstetrics because the few available studies are retrospective, all have small numbers of patients, and the studies have given conflicting results regarding the safety of retaining a cerclage after preterm premature rupture of the membranes. It is unclear from the retrospective studies whether latency (the interval from membrane rupture to the onset of labor) is prolonged with retention of the suture. Furthermore, some, but not all studies suggest an increase in major infectious maternal morbidity and possibly neonatal morbidity. For this reason, clinicians vary greatly in deciding on whether to remove a cerclage in a patient with PPROM and either practice is currently an acceptable standard. This is a fairly rare complication, the combination of PPROM in a patient with cerclage in place only occurs in about 1-3/1000 pregnant women. Thus it has been impossible to study this problem prospectively in any single institution. The establishment of the Obstetrix Collaborative Research Group affords the unique opportunity to study this rare complication. Obstetrix manages 19 practices of Perinatologists around the U.S. and Mexico and is comprised of nearly 100 such subspecialists. This problem is most often referred to a Perinatologist when it occurs, so it is not unusual for these practices to see 5 - 10 such patients per year. Obstetrix fully funds the infrastructure of this research group and inclusion in this study will not alter the cost of patient care in either group as there is virtually no cost in removing the cerclage and all these patients are kept in hospital until delivery when membranes rupture as standard of care.

This is a multicenter trial. The purpose is to determine whether retention of cerclage after preterm premature rupture of the membranes improves latency (without a significant increase in chorioamnionitis) and lessens neonatal morbidity.

ELIGIBILITY:
Inclusion Criteria:

1. A previously placed prophylactic cerclage defined as any cerclage done < 23 6/7 weeks including those done for previous history of cervical incompetence, asymptomatic cervical shortening (regardless of effacement) and asymptomatic cervical dilation < 3 cm
2. Spontaneous rupture of membranes 22-32 weeks
3. Singleton or twin gestation
4. Shirodkar or McDonald cerclage in place > 1 week

Exclusion Criteria:

1. Active labor (> 8 uterine contractions [UCs] per hour)
2. Chorioamnionitis as defined by temperature > 38 plus fetal tachycardia or uterine tenderness
3. Placenta previa or undiagnosed vaginal bleeding
4. Nonreassuring fetal status by nonstress test (NST) or biophysical profile (BPP)
5. Mature pulmonary studies
6. Positive gram stain, culture, white blood cells (WBC) > 30, or glucose < 14 on amniocentesis
7. Major fetal anomaly
8. Presentation > 48 hours after rupture of membranes
9. abdominal cerclage
10. Cerclage done for symptomatic cervical dilation (cervix dilated > 3 cm)
11. Post amniocentesis membrane rupture (rupture which occurs within one week of amniocentesis)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2004-11; Primary Completion 2013-11 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Chorioamnionitis as defined by temperature > 38 plus fetal tachycardia or uterine tenderness | conception to birth
Composite neonatal outcome - any one of the following (for twins, either infant): Fetal or neonatal death | Birth to 28days of life
Respiratory distress syndrome | birth to 28days of life
Documented sepsis within 72 hours of delivery | birth to 72 hours after delivery
Grade 3 or 4 intraventricular hemorrhage | birth to 28days of life
Stage 2 or 3 necrotizing enterocolitis | birth to 28days of life
Neonatal intensive care unit (NICU) stay | birth to 28days of life
Birth weight | at birth
Estimated gestational age (EGA) at delivery | at delivery
Postpartum endometritis | birth to 28days of life
Maternal sepsis | birth to 28days following delivery
Latency | labor to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Maurel, RN, MSN, CNS, Study Director — Obstetrix Medical Group, Inc.
Locations (23):
- United States (23):
  - Desert Good Samaritan Hospital, Mesa, Arizona
  - Banner Good Samaritan Hospital, Phoenix, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - Saddleback Memorial Medical Center, Laguna Hills, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - University of Southern California-Irvine Medical Center, Orange, California
  - Good Samaritan Hospital, San Jose, California
  - Swedish Medical Center, Denver, Colorado
  - Presbyterian/St Luke's Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Yale New-Haven Medical Center, New Haven, Connecticut
  - University of Illinois at Chicago, Chicago, Illinois
  - Lousiana State University Health Science, Shreveport, Louisiana
  - Hutzel Women's Hospital, Detroit, Michigan
  - Saint Luke's Hospital, Kansas City, Kansas City, Missouri
  - Sunrise Medical Center, Las Vegas, Nevada
  - University of Rochester Medical Center, Rochester, New York
  - The University Hospital, Cincinnati, Ohio
  - Sacred Heart Medical Center, Eugene, Oregon
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Memorial Hermann Children's Hospital-Texas Center for Fetal Assessment, Houston, Texas
  - Evergreen Hospital, Kirkland, Washington
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Background] Treadwell MC, Bronsteen RA, Bottoms SF. Prognostic factors and complication rates for cervical cerclage: a review of 482 cases. Am J Obstet Gynecol. 1991 Sep;165(3):555-8. doi: 10.1016/0002-9378(91)90283-w. PMID 1892180
- [Background] American College of Obstetricians and Gynecologists. Preterm Labor. Technical Bulletin no. 206,1995.
- [Background] McElrath TF, Norwitz ER, Lieberman ES, Heffner LJ. Management of cervical cerclage and preterm premature rupture of the membranes: should the stitch be removed? Am J Obstet Gynecol. 2000 Oct;183(4):840-6. doi: 10.1067/mob.2000.108870. PMID 11035323
- [Background] Jenkins TM, Berghella V, Shlossman PA, McIntyre CJ, Maas BD, Pollock MA, Wapner RJ. Timing of cerclage removal after preterm premature rupture of membranes: maternal and neonatal outcomes. Am J Obstet Gynecol. 2000 Oct;183(4):847-52. doi: 10.1067/mob.2000.109039. PMID 11035324
- [Background] Ludmir J, Bader T, Chen L, Lindenbaum C, Wong G. Poor perinatal outcome associated with retained cerclage in patients with premature rupture of membranes. Obstet Gynecol. 1994 Nov;84(5):823-6. PMID 7936520
- [Background] Naylor CS, Gregory K, Hobel C. Premature rupture of the membranes: an evidence-based approach to clinical care. Am J Perinatol. 2001 Nov;18(7):397-413. doi: 10.1055/s-2001-18699. PMID 11731894
- [Derived] Galyean A, Garite TJ, Maurel K, Abril D, Adair CD, Browne P, Combs CA, How H, Iriye BK, Kominiarek M, Lu G, Luthy D, Miller H, Nageotte M, Ozcan T, Porto M, Ramirez M, Sawai S, Sorokin Y; Obstetrix Perinatal Collaborative Research Network. Removal versus retention of cerclage in preterm premature rupture of membranes: a randomized controlled trial. Am J Obstet Gynecol. 2014 Oct;211(4):399.e1-7. doi: 10.1016/j.ajog.2014.04.009. Epub 2014 Apr 12. PMID 24726507